CLINICAL TRIAL: NCT04168502
Title: Phase 3 Study to Assess Gemtuzumab, in Combination With Standard Chemotherapy, on MRD Levels, in Adult, 18-60 Years, With Previously Untreated de Novo Fav-interm Risk AML
Brief Title: Gemtuzumab Chemotherapy MRD Levels; Adult Untreated, de Novo, Fav Interm Risk AML
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML1819
Record Dates: First submitted 2019-11-11; First posted 2019-11-19 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: De-novo; Favorable risk; Intermediate risk; Gemtuzumab ozogamicin; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Induction:
  Gemtuzumab 3 mg/m2 day 1,4,7 Daunorubicin 60 mg/m2 day 1-3 Cytosine arabinoside 200 mg/m2 day 1-7
  Consolidation:
  Gemtuzumab 3 mg/m2 day 1 Daunorubicin 50 mg/m2 day 4-6 Cytosine arabinoside 500 mg/m2 twice a day, day 1-6
  Allogeneic transplantation or Autologous transplantation according to MRD level
  clinical observation
  Interventions: Drug: Gemtuzumab Ozogamicin

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin — Patients will receive induction and consolidation with Gemtuzumab ozogamicin, Daunorubicin and Cytarabine

SUMMARY:
MRD driven study. Addition of gemtuzumab to conventional chemotherapy to reduce MRD of patients with favorable/intermediate-risk AML. Post-consolidation assessment of MRD.

DETAILED DESCRIPTION:
Setting up a multicenter, MRD (Minimal Residual Disease)-driven study that relies on addition of gemtuzumab ozogamicin to conventional chemotherapy to reduce the pre-transplant levels of MRD of patients with favorable/intermediate-risk (according to ELN 2017) AML. Post-consolidation assessment of MRD will be exploited to establish the final risk assignment and to verify whether the delivery of a post remission therapy intensity (AuSCT, Autologous Stem Cell Transplant, vs ASCT, Allogeneic Stem Cell Transplant) of which is MRD-driven will improve the outcome in terms of anti-leukemic efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent according to ICH/EU/GCP and national/local laws
2. Patients aged between 18 and 60 years
3. Patients previously untreated for their AML by other chemotherapeutic agents (except for no more than 7 days HU) or radiotherapy
4. Unequivocal diagnosis of de novo AML according to WHO diagnostic criteria (at least 20% blasts in the bone marrow), other than acute promyelocytic leukemia, documented by bone marrow aspiration (or biopsy in case of dry tap) (not supervening after other myeloproliferative disease or myelodysplastic syndromes of ≥ 6 months duration)
5. Patients with favorable-intermediate AML according to ELN 2017 (except for FLT3-ITD/TKD positive AML)
6. WHO performance status 0-3
7. Adequate renal (serum creatinine ≤ 2 x the institutional ULN) and liver (total serum bilirubin ≤ 2 x ULN; serum ALT and AST ≤ 2.5 x ULN) function, unless considered due to organ leukemic involvement
8. Left Ventricular Ejection Fraction (LVEF) ≥ 50%, as determined by echocardiogram
9. Absence of severe concomitant neurological or psychiatric diseases and congestive heart failure or active uncontrolled infection
10. Absence of any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and the follow-up schedule.

Exclusion Criteria:

1. Patients already treated for their AML by other chemotherapeutic agents (except for no more than 7 days HU) or radiotherapy
2. Acute promyelocytic leukemia
3. Blast crisis of chronic myeloid leukemia
4. FLT3-ITD/TKD positive AML
5. AML supervening after other myeloproliferative disease
6. AML supervening after antecedent myelodysplastic syndromes ≥ 6 months duration
7. Therapy-related AML
8. Other active or progressive malignant diseases.
9. Inadequate renal or liver function (metabolic abnormalities > 2-2.5 times the normal upper limit)
10. Severe heart failure requiring diuretics
11. Ejection fraction < 50%
12. Uncontrolled infections
13. Severe concomitant neurological or psychiatric diseases
14. Patients who are pregnant or adults of reproductive potential not employing an effective method of birth control. Women of childbearing potential must have a negative serum pregnancy test within 48 hours prior to administration of chemotherapy. Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients must agree to employ an effective barrier method of birth control throughout the study and for at least 6 months following discontinuation of study drug.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 414 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Activity of GO in combination with chemotherapy in terms of MRD negativity achievement | 2 months
  Percentage of MRD negativity after consolidation in patients treated in induction and consolidation with GO

CONTACTS AND LOCATIONS:
Locations (48):
- Italy (48):
  - A.O. - SS. Antonio e Biagio e Cesare Arrigo - SC Ematologia, Alessandria
  - Aou Ospedali Riuniti "Umberto I - G.M. Lancisi - G. Salesi"- Ancona - Sod Clinica Ematologica, Ancona
  - Area Vasta N. 5 Ascoli Piceno - S. Benedetto Del Tronto, Presidio Ospedaliero Av5 Osp. Gen. Prov.Le "C.G.Mazzoni" - Uoc Ematologia, Ascoli Piceno
  - AO "San Giuseppe Moscati" - UOC Ematologia con unità di trapianto, Avellino
  - AOU Consorziale Policlinico "Aldo Moro" - UO Ematologia con trapianto, Bari
  - Policlinico S. Orsola - Malpighi - UOC Ematologia, Bologna
  - Ao Sant'Anna E San Sebastiano - Caserta - Uoc Onco Ematologia, Caserta
  - U.O.C. Oncoematologia - Istituto Oncologico Veneto Irccs, Presidio Ospedaliero S. Giacomo Apostolo, Castelfranco Veneto
  - Asur Marche Area Vasta 3 - Presidio Ospedaliero Civitanova Marche - Uods Ematologia, Civitanova Marche
  - Aou Arcispedale Sant'Anna - Cona (Fe) - Uoc Ematologia E Fisiopatologia Della Coagulazione, Cona
  - Asst Di Cremona - Ospedale Di Cremona - Uo Ematologia, Cremona
  - Aou Careggi - Firenze - Sod Ematologia, Florence
  - Asl Frosinone, Ospedale F. Spaziani - Ematologia, Frosinone
  - Irccs Aou San Martino - Genova - Uo Ematologia E Trapianti, Genova
  - Presidio Ospedaliero Nord "Santa Maria Goretti" - UOC Ematologia, Latina
  - ASL Le/1 P.O. Vito Fazzi - UO Ematologia, Lecce
  - Aulss 3 Serenissima, Ospedale Dell'Angelo - Mestre - Uo Ematologia, Mestre
  - Asst Grande Ospedale Metropolitano Niguarda - Milano - Sc Ematologia, Milan
  - Irccs Ospedale S. Raffaele - Milano - Uo Oncoematologia, Milan
  - ISTITUTO EUROPEO DI ONCOLOGIA IRCCS - MILANO - DIVISIONE DI ONCOEMATOLOGIA 176 Milano Divisione di Onco-Ematologia Istituto Europeo, Milan
  - Aou Di Modena - Sc Ematologia, Modena
  - Ao Di Rilievo Nazionale Antonio Cardarelli - Napoli - Uoc Ematologia Con Trapianto Di Midollo, Napoli
  - Aou Federico Ii - Napoli - Uoc Ematologia, Napoli
  - Aou San Luigi Gonzaga - Orbassano - Scdu Ematologia Generale E Oncoematologia, Orbassano
  - Asl Salerno, Presidio Ospedaliero Tortora Pagani - Ematologia, Pagani
  - Ao Ospedali Riuniti Villa Sofia Cervello - Palermo - Uo Ematologia Con Utmo, Palermo
  - Aou Policlinico P. Giaccone - Palermo - Uo Ematologia, Palermo
  - Fondazione Ircss Policlinico San Matteo - Pavia - Uo Ematologia, Pavia
  - Ao Di Perugia, Ospedale S. Maria Della Misericordia - Ematologia E Trapianto Midollo Osseo, Perugia
  - Ao Ospedali Riuniti Marche Nord - Ospedale San Salvatore - Pesaro - Uoc Ematologia E Centro Trapianti, Pesaro
  - Asl Pescara, Presidio Ospedaliero 'Spirito Santo' - Uoc Ematologia Clinica, Pescara
  - Asl Di Piacenza, Ospedale "Guglielmo Da Saliceto" - Ematologia E Centro Trapianti, Piacenza
  - Ausl Della Romagna, Ospedale "Santa Maria Delle Croci" - Ravenna - Ematologia, Ravenna
  - Ausl Di Reggio Emilia - Arcispedale Santa Maria Nuova, Irccs - Sc Ematologia, Reggio Emilia
  - Ausl Della Romagna, Ospedale "Infermi" - Rimini - Uo Ematologia, Rimini
  - Ao Complesso Ospedaliero San Giovanni / Addolorata - Roma - Uoc Ematologia, Roma
  - AOU Policlinico Tor Vergata- UOC Trapianto cellule staminali, Roma
  - Aou Sant'Andrea - Roma - Uoc Ematologia, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs - Roma - Area Ematologica, Roma
  - Istituti Fisioterapici Ospitalieri - Ifo - Istituto Regina Elena - Roma - Uosd Ematologia, Roma
  - Policlinico Universitario Campus Bio Medico - Roma - Uoc Ematologia E Trapianto Di Cellule Staminali, Roma
  - Università Degli Studi Di Roma "Sapienza" - Dipartimento Di Medicina Traslazionale E Di Precisione - U.O.C. Ematologia, Roma
  - Ente Ecclesiastico Casa Sollievo Della Sofferenza - San Giovanni Rotondo - Ematologia, San Giovanni Rotondo
  - Aou Di Sassari - Cliniche Universitarie - Stabilimento Cliniche Di San Pietro - Uoc Ematologia, Sassari
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia 2, Torino
  - Unità Operativa Di Ematologia - Presidio Ospedaliero Di Treviso - Azienda Ulss N.2 Marca Trevigiana, Treviso
  - Azienda Sanitaria Universitaria Integrata Di Trieste - Sc Ematologia, Trieste
  - Asui Di Udine - Presidio Ospedaliero "Santa Maria Della Misericordia" - Clinica Ematologica, Udine